CLINICAL TRIAL: NCT05625672
Title: EVALUATION OF THE EFFICIENCY OF HEMOVIGILANCE MODULE TRAININGS
Brief Title: EFFICIENCY OF HEMOVIGILANCE MODULE TRAININGS GIVEN TO NURSES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-38
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Nurse's Role; Training Group, Sensitivity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Randomized, parallel-group, placebo-controlled study
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Five modules of training on hemovigilance were given in 5 hours. A pre-test was applied at the beginning of the training. The final test was done at the end of the training. One month later, the same test was applied again to measure the permanence of the training.
  Interventions: Other: Training
- Control (No Intervention): No training was provided. Only the pretest was administered one week after the posttest.

INTERVENTIONS:
Other: Training — Hemovigilance module training
  Arms: Intervention

SUMMARY:
The aim of the present study is to determine the effectiveness of hemovigilance module training given to nurses.

DETAILED DESCRIPTION:
125 nurses from the clinic and intensive care units, who received the most intensive blood transfusion from two different hospitals, were included in the study as the intervention and control groups. The control group was not trained. Only the pretest was administered one week after the posttest. After the pre-test was applied to the nurses in the intervention group, five modules of training, which lasted four hours, were given using interactive methods. Five modules of training were prepared by the researcher. These five modules are the 1st module of training; definition of hemovigilance, its aims, the development of hemovigilance in the world and in Turkey, and legal legislation, Module 2; Donor selection, Blood donation Process, Phlebotomy and Donor reactions, Module 3; blood, blood transfusion, its purpose, properties of blood and blood components, Blood transfusion process, Module 4; acute and delayed transfusion reactions and management, Module 5; It consists of the national hemovigilance system, the organization of the hemovigilance system at the hospital level, Traceability, Trace-back from the Patient to the Donor, and Look-back from the Donor to the Patient. the training was over, the final test was administered. One month later, this test was repeated.

ELIGIBILITY:
Inclusion Criteria:

She/He voluntarily agrees to participate in the research, Working as a nurse in the clinic and intensive care unit where blood transfusions are the most, Working for at least 6 months,

Exclusion Criteria:

Nurses working in the emergency and operating rooms, in clinics where blood transfusion is not performed the most, Being a new nurse, On maternity leave and maternity leave, Having an external assignment, Nurses working in the polyclinic,

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Hemovigilance Information Form | 5 hours or 1 month
  It consists of fifteen questions about hemovigilance and hemovigilance system and definitions.
Information Form on Blood Transfusion Complications | 5 hours or 1 month
  This section consists of nine questions including transfusion complications.
Information Form on Blood Transfusion Applications | 5 hours or 1 month
  This section consists of sixteen questions including donor selection, questions about blood components, blood group and safe blood transfusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No